CLINICAL TRIAL: NCT02733302
Title: Hope Theory as Ability Determinant to Permanently Change the Adapted Physical Activity (APA) in Type 2 Diabetic Patients
Acronym: APADIAB-ESPOIR
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2015-A01815-44
Record Dates: First submitted 2016-03-30; First posted 2016-04-11 (Estimated); Last update posted 2017-11-01 (Actual); Status verified 2017-10

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Hope theory (Experimental)
  Interventions: Behavioral: Hope theory

INTERVENTIONS:
Behavioral: Hope theory — Adapted Physical Activity

SUMMARY:
The control of diabetes is related both to food, treatment but also to physical activity. Despite these recommendations and these positive findings, patients are always sedentary because of brakes in the practice of a regular physical activity.

It is therefore interesting to consider the representations of patients and particularly on the way of establishment in order to reach a goal. The Hope Theory highlights the hope as the sum of the will and means that an individual has to achieve its goals. Will be discussed in this study to identify a relationship between the level of hope for patients and their ability to permanently change their behavior in regular physical activity as part of the goals set during the week of therapeutic education patient.

ELIGIBILITY:
Inclusion Criteria:

* Major Topic
* Type 2 Diabetic Topic
* Inactive Topic
* Subject of CHU ANGERS hospitalized for a week Diab'Equilibre, Diabetology Service
* Subject participating in the service of the APA program
* Subject who understands and reads French
* Subject has given its consent to participate signed the protocol

Exclusion Criteria:

* Removing the participation of consent;
* Severe heart failure
* Severe respiratory failure
* Bone metastases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2016-04-04 (Actual); Primary Completion 2019-08 (Estimated); Study Completion 2019-09 (Estimated)

PRIMARY OUTCOMES:
IPAQ-SF questionnaire for measure of Physical Activity | 6 month

CONTACTS AND LOCATIONS:
Locations (1):
- UHAngers, Angers, France